CLINICAL TRIAL: NCT03277586
Title: Effects of Probiotics on Symptoms of Depression
Acronym: EPSD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Dr. Roumen Milev (Other)
Responsible Party: Sponsor-Investigator, Dr. Roumen Milev, Head, Department of Psychiatry, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6020656
Record Dates: First submitted 2017-09-01; First posted 2017-09-11 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2021-01

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 16-week Double-blind randomized placebo-controlled dual-phase trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probio'Stick (Experimental)
  Interventions: Drug: Probio'Stick
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probio'Stick — Probiotic supplement containing Lactobacillus helveticus and Bifidobacterium longum
  Arms: Probio'Stick
Drug: Placebo — Identically formulated and packaged inactive substance
  Arms: Placebo

SUMMARY:
Preclinical and clinical studies have shown that consuming probiotics can improve mood, anxiety, and cognition, as well as alter brain activity in both rodents and healthy humans. Data from our recent open-label, 8-week pilot study provided the first evidence of these effects in depressed patients, with significant improvements observed in overall mood, anhedonia, and sleep quality. To further support this evidence and expand upon the search for biomarkers in depression, data from this pilot study is being used to plan a 16-week, double-blind randomized placebo-controlled trial to assess the effects of probiotics on depression. Participants diagnosed with depression recruited from the greater Kingston area will orally consume a probiotic supplement containing Lactobacillus helveticus and Bifidobacterium longum (Probio'Stick, Lallemand Health Solutions) or placebo once daily. Participants will undergo clinical assessments measuring mood, anxiety, cognition, and sleep using a battery of validated clinical scales to assess efficacy of the probiotic alleviating depressive symptoms; sleep will also be assessed objectively with an ambulatory polysomnogram. Neuroimaging data will be collected using magnetic resonance imaging and electroencephalography to look at functional, structural, and electrical changes in the brain associated with consumption of the probiotic. Molecular data will be collected from blood, stool, and urine samples to look at levels of cytokines and serotonin, and explore potential genes and proteins that may predict outcomes in depression. An informatics-based approach will be used to integrate clinical, neuroimaging, and molecular data to look for biomarkers that indicate disease state and predict antidepressant-like response to the probiotic. Results: We expect results to replicate and expand on our pilot data, demonstrating that probiotics are effective in alleviating symptoms of depression, and to find biomarkers that will predict these outcomes. The findings from this study will contribute robust scientific data that is currently lacking in this emerging field.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Major Depressive Disorder (MDD) according to DSM-5 as determined by MINI
2. Current depressive episode with a MADRS score of 20
3. Males and females between ages 18 and 65
4. Able to understand and comply with the requirements of the study
5. Provision of written informed consent

Exclusion Criteria:

1. Current use of any antidepressant drug
2. Three or more previous episodes of depression
3. Failure to respond to another treatment in the current episode
4. Use of any antibiotic drug in the past 4 weeks (may be eligible to participate after a 1-month washout period). Should a participant require an antibiotic drug during the 16 week study period, they may continue with the study but must take the probiotic 4-6 hours before or after they take the antibiotic.
5. Use of any sleep medication in the past 4 weeks (may be eligible to participate after a 1-month washout period)
6. Milk, yeast, or soy allergy
7. History of alcohol or substance dependence in the past 6 months
8. Use of probiotic product in the past 2 weeks (may be eligible to participate after a 2-week washout period) and during the trial
9. Use of any type of laxative
10. Consumption of products fortified in probiotics 2 weeks before and during the trial
11. High risk of suicide (score 4 or more on item 10 of MADRS)
12. Psychotic symptoms determined by the MINI
13. Bipolar Disorder determined by the MINI
14. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial (determined by a pregnancy test performed at the screening visit and confirmation of the use of appropriate contraception)
15. Immunodeficiency (immuno-compromised and immuno-suppressed participants; e.g. AIDS, lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participants)
16. Unstable or severe medical conditions (e.g. cancer, cardiovascular, renal, lung, diabetes, psychiatric illness, bleeding disorders, etc.)
17. The use of natural health products (NHPs; e.g. St. John's Wort, melatonin, passion flower, etc.) that affect depression or sleep is not allowed in the trial
18. Electroconvulsive therapy (ECT) in the year prior to participation in the study
19. Taking medication or other not-permitted treatment that cannot be safely discontinued

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Mood | 16 weeks
  Montgomery-Asberg Depression Rating Scale

SECONDARY OUTCOMES:
Anxiety | 16 weeks
  Generalized Anxiety Disorder 7-item Scale
Anhedonia | 16 weeks
  Snaith Hamilton Pleasure Scale
Cognition | 16 weeks
  CNS Vital Signs
Cytokines | 16 weeks
  Blood plasma
Serotonin | 16 weeks
  Blood Plasma
Microbiome | 16 weeks
  Stool
Brain structure/function | 8 weeks
  fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No